CLINICAL TRIAL: NCT04825808
Title: Detailed Clinical and MRI Characteristics in Primary Non-traumatic Convexity Subarachnoid Haemorrhage Elderly Patients.
Acronym: cSAH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2021/DR-01
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Amyloid Angiopathy; Subarachnoid Hemorrhage
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Consecutive elderly (≥55 years) patients, recruited and registered in the stroke database of two centres (Nîmes University Hospital and Montpellier University Hospital, France), presenting with cSAH with suspected, possible, or probable CAA.
  Interventions: Other: usual care

INTERVENTIONS:
Other: usual care — according to recommendations

SUMMARY:
Transient focal neurological episode (TFNE) is the most frequent presenting symptom of convexity subarachnoid haemorrhage (cSAH) in elderly patients with non-traumatic cSAH with suspected, possible or probable cerebral amyloid angiopathy (CAA). The aim of our study was to analyse in detail clinical and MRI characteristics in these patients.

Methods: We performed a retrospective study analysing baseline, acute clinical symptom (TFNE and headache), and MRI characteristics (acute cSAH and chronic CAA features) of consecutive elderly (≥55 years) patients, recruited and registered in the stroke database, between june 2008 and october 2020 of two centres (Nîmes and Montpellier University Hospital, France), presenting with cSAH with suspected, possible, or probable CAA.

ELIGIBILITY:
Inclusion Criteria:

* ≥55 years of age,
* acute symptomatic cSAH based on FLAIR and T2*-weighted imaging performed within one month of symptom onset, recent trauma,
* anticoagulation treatment, pathological blood coagulation tests (activated partial thromboplastin time [aPTT] ratio=patient's aPTT/normal control aPTT] >1.2; or partial thromboplastin time [PTT] <75%) or platelet count (<100 x 109/L),

Exclusion Criteria:

* exclusion of underlying non-CAA cSAH causes (e.g. reversible cerebral vasoconstriction syndrome, trauma, cerebral venous sinus thrombosus, aneurysm, primary angiitis of the central nervous system, anticoagulation treatment, pathological blood coagulation tests)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive elderly (≥55 years) patients, recruited and registered in the stroke database of two centres (Nîmes University Hospital and Montpellier University Hospital, France), presenting with cSAH with suspected, possible, or probable CAA.
  The patients were classified as possible or probable CAA according to the modified Boston criteria. Since cortical superficial siderosis (CSS), incorporated in the modified Boston criteria, is probable a result of an earlier acute cSAH, we considered patients with acute cSAH in the absence of other typical CAA-related haemorragic features as patients with suspected CAA.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Description of MRI | day of the diagnosis
  Extent of acute cSAH (number of sulci, focal [≤3 sulci] or diffuse [>3 sulci], surface)
Description of MRI | day of the diagnosis
  the multifocality of acute cSAH (as described for cortical superficial siderosis (CSS)), sulci involved by cSAH, CSS presence, CSS extent (focal, ≤3 sulci; diffuse >3 sulci)
Description of MRI | day of the diagnosis
  cerebral microbleeds (CMB, <10 mm) presence
Description of MRI | day of the diagnosis
  cerebral microbleeds number
Description of MRI | day of the diagnosis
  cerebral microbleeds categorisation (according to the Microbleed Anatomical Rating Scale),
Description of MRI | day of the diagnosis
  presence and number of chronic lobar intracerebral haemorrhage (ICH) (>10 mm)
Description of MRI | day of the diagnosis
  Extent of white matter hyperintensities (periventricular Fazekas scale 0-3)
Clinical parameters | day of the diagnosis
  Transient focal neurological episode (TFNE) presence
Clinical parameters | day of the diagnosis
  number of TFNE preceding MRI
Clinical parameters | day of the diagnosis
  TFNE symptoms (sensory, motor, visual, speech; positive or negative symptoms
Clinical parameters | day of the diagnosis
  Presence and speed of spreading TFNE symptoms
Clinical parameters | day of the diagnosis
  Correlation of TFNE symptoms to cSAH localisation
Clinical parameters | day of the diagnosis
  headache (Yes/No)
Clinical parameters | day of the diagnosis
  antiepileptic drugs (AED) introduction and type of AED introduced

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Derived] Autieri V, Gaillard N, Mourand I, Laurent-Chabalier S, Mura T, Trandafir C, Wacongne A, de Champfleur NM, Thouvenot E, Pereira F, Renard D. Primary acute convexity subarachnoid hemorrhage in older patients: analysis of baseline, clinical and MRI characteristics including quantitative surface study and topographical probabilistic mapping of convexity subarachnoid hemorrhage. Acta Neurol Belg. 2023 Apr;123(2):519-527. doi: 10.1007/s13760-022-02115-8. Epub 2022 Oct 14. PMID 36241843